CLINICAL TRIAL: NCT02584647
Title: Phase I Study Evaluating Combination Therapy With the Receptor Tyrosine Kinase Inhibitor PLX3397 and Sirolimus in Patients With Unresectable Sarcoma and Phase II Study in Malignant Peripheral Nerve Sheath Tumors
Brief Title: PLX3397 Plus Sirolimus in Unresectable Sarcoma and Malignant Peripheral Nerve Sheath Tumors
Acronym: PLX3397
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Gulam Manji (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor-Investigator, Gulam Manji, Assistant Professor of Medicine (Oncology), Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAO6059; R01FD005745 (FDA)
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Sarcoma; Malignant Peripheral Nerve Sheath Tumors
Keywords: Unresectable
MeSH Terms: conditions — Sarcoma; Neurofibrosarcoma | interventions — pexidartinib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: PLX3397 and Sirolimus (Experimental): Subjects with unresectable or metastatic sarcoma will take orally PLX3397 (600 - 1000mg) in combination with Sirolimus (2-6mg) daily.
  Interventions: Drug: PLX3397; Drug: sirolimus
- Phase 2: PLX3397 and Sirolimus (Experimental): Subjects with unresectable or metastatic Malignant Peripheral Nerve Sheath Tumors (MPNSTs) will take PLX3397 and Sirolimus at the recommended Phase 2 dose (RP2D).
  Interventions: Drug: PLX3397; Drug: sirolimus

INTERVENTIONS:
Drug: PLX3397 — PLX3397 is a small molecule that potently and selectively inhibits macrophage colony-stimulating factor receptor (FMS), Kit, and FMS-like tyrosine kinase 3 (Flt3)-internal tandem duplication (ITD) kinases, which regulate key components of the tumor microenvironment and oncogenic variants of these kinases that drive certain tumors.
  Other Names: pexidartinib
Drug: sirolimus — Sirolimus is a macrocyclic lactone that binds to tacrolimus (FK506) binding protein 12 and inhibits mammalian target of rapamycin (mTOR) resulting in cell-cycle arrest and apoptosis.
  Sirolimus is currently approved as an immunosuppressive agent for organ transplantation and more recently, as a component of cardiac arterial stents because of its potent antiproliferative effects on fibroblasts responsible for restenosis after such a procedure (26) Sirolimus is commonly administered orally on a daily basis, in doses ranging from 2 to 40 mg/day.
  Other Names: Rapamune

SUMMARY:
The purpose of this study is to determine if treatment with PLX3397 and Sirolimus will be tolerated and result in shrinking of the cancer or stopping the cancer from growing. In the phase I portion, the maximum tolerate dose of the study drug will be determined. In the Phase II portion, progression free survival will be assessed at the dose level found in Phase I. Participants will continue to take the study drug until they experience an unacceptable side effect or their disease progresses. Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Malignant peripheral nerve sheath tumors (MPNSTs) represent up to 10% of adult soft tissue sarcomas. Due to its rarity, few MPNST-specific prospective trials exist, and treatments are largely based on extrapolation from results from other sarcoma subtypes. Since the molecular pathways driving pathogenesis within sarcoma subtypes are distinct, these treatment options are likely suboptimal at best. Targeted therapies that block key pathways known to drive MPNST will likely result in superior tumor responses with limited toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Disease site/type with pathologic confirmation of diagnosis at participating cancer site.

  * Phase 1: Advanced, unresectable sarcoma (any subtype)
  * Phase 2: Advanced, unresectable malignant peripheral nerve sheath tumors (MPNSTs)
* Extent of disease: Unresectable
* Allowable prior therapy

  * Phase 1: Progressed on standard of care therapy with up to three prior treatments
  * Phase 2: MPNST with 0-3 prior systemic treatments (no prior radiotherapy is necessary).
* Eastern Cooperative Oncology Group (ECOG) performance status: 0, 1, or 2
* Age greater or equal to 18 years. Because no dosing or adverse event data are currently available on the use of PLX3397 in combination with sirolimus in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Presence of measurable lesions by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Allowable laboratory values with date range

  * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L, hemoglobin (Hgb) >9 g/dL, and platelet count ≥100 X 10^9/L
  * Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ upper limit of normal (ULN) or < 2.5 x ULN in the presence of liver metastases, bilirubin ≤ 1.5 x ULN, albumin ≥ 3.0g/dL.
  * Bilirubin ≤ ULN; patients with hyperbilirubinemia clinically consistent with an inherited disorder of bilirubin metabolism (e.g., Gilbert syndrome) will be eligible at the discretion of the principal investigator.
  * Albumin ≥ 3.0g/dL.
  * Creatinine ≤ 1.5 x ULN or calculated creatinine clearance (CrCl) > 60 mL/min using the Cockcroft-Gault formula less than eight days pior to start of treatment.
* Women of child-bearing potential must have a negative serum pregnancy test at screening and must agree to use an effective form of contraception from the time of the negative pregnancy test and for a minimum of 3 months after the last dose of study drug. Effective forms of contraception include abstinence, hormonal contraceptive (injectable or implantable) in conjunction with a barrier method, or a double barrier method. Women of non-child-bearing potential must have been postmenopausal for ≥ 1 year or surgically sterile. The effects of PLX3397 and sirolimus on the developing human fetus are unknown. For this reason women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after completion of PLX3397 and sirolimus administration.
* Fertile men must agree to use an effective method of birth control during the study and for up to 3 months after the last dose of study drug.
* Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements.
* Agree to pre and post-treatment tumor biopsies.
* Prior treatment-related Adverse Events must be ≤ grade 1 (CTCAE v4.0), except alopecia, at time of initiating study drug.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier or within 14 days from cycle 1 day 1 of PLX3397 and sirolimus.
* Patients who are receiving any other investigational agents concurrently.
* Concomitant treatment with other anti-neoplastic agents (hormonal therapy acceptable).
* Patients with symptomatic brain metastases. Subjects with untreated brain metastasis ≤ 1 cm can be considered eligible if deemed asymptomatic by the investigator upon consultation with the medical monitor and do not require immediate radiation or steroids. Subjects with brain metastasis that is treated and stable for 1 month may be considered eligible if they are asymptomatic and on stable dose of steroids or if they do not require steroids following successful local therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PLX3397 or sirolimus.
* For Phase 2 - Prior exposure to a receptor tyrosine kinase or mammalian target of Rapamycin inhibitor.
* Pregnant women are excluded from this study because PLX3397 and sirolimus are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with PLX3397 and sirolimus, breastfeeding should be discontinued if the mother is treated with PLX3397 and sirolimus.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active liver disease, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active secondary malignancy unless the malignancy is not expected to interfere with the evaluation of safety and is approved by the Sponsor. Examples of the latter include basal or squamous cell carcinoma of the skin, in-situ carcinoma of the cervix, and isolated elevation of prostate-specific antigen. Subjects with a completely treated prior malignancy and no evidence of disease for ≥ 2 years are eligible.
* Major surgical procedure or significant traumatic injury within 14 days of initiating study drug or anticipation of the need for major surgery during the study.
* Previous radiotherapy to 25% or more of the bone marrow and/or radiation therapy within 28 days prior to study entry.
* Inability to swallow capsules, or refractory nausea and vomiting, malabsorption, an external biliary shunt, or significant bowel resection that would preclude adequate absorption.
* Congestive heart failure (CHF) New York (NY) Heart Association class III or IV; unstable coronary artery disease (myocardial infarction (MI) more than 6 months prior to study entry is permitted); or serious cardiac arrhythmia.
* Baseline QTc corrected by Fridericia's formula (QTcF) ≥ 450 ms (males) or ≥ 470 ms (females)
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with PLX3397. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Similarly, patients with chronic or acute hepatitis C virus (HCV) or hepatitis B virus (HBV) infection are also ineligible.
* Of the five major cytochrome P450 (CYP) isoforms, 3A4 (BFC) may be involved in Phase I metabolism of PLX3397, with possibly CYP1A2 playing a minor role. Until information regarding exposure toxicity and exposure-response relationships are available with PLX3397, concomitant strong CYP3A4 inhibitors and inducers are not permitted in the event they alter the systemic exposure to PLX3397 (see Attachment 1 for a list of common CYP3A4 inhibitors and inducers). These include anticonvulsants, mycin antimicrobials, and antiretrovirals. Some common examples include inhibitors such as erythromycin, fluoxetine, gemfibrozil, and inducers such as rifampicin, carbamazepine, phenytoin, efavirenz, and nevirapine. Concomitant treatment is permitted if the medication is not expected to interfere with the evaluation of safety or efficacy of the study drug. Sirolimus undergoes extensive hepatic and intestinal metabolism via CYP3A4 and CYP3A5, as well as excretion by P-glycoprotein. Strong CYP3A inhibitors such as ketoconazole or grapefruit juice are not permitted. Patients should be monitored for supratherapeutic toxic levels of sirolimus and PLX3397. As bone marrow suppression including anemia, neutropenia, and thrombocytopenia have been reported in patients receiving sirolimus monotherapy, these adverse effects may be exacerbated in combination with PLX3397 for which patients will be closely monitored.
* Any patients on warfarin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2023-07 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gulam A. Manji, MD, Principal Investigator — Columbia University
Locations (5):
- United States (5):
  - University of Iowa, Iowa City, Iowa
  - Early Drug Development Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manji GA, Van Tine BA, Lee SM, Raufi AG, Pellicciotta I, Hirbe AC, Pradhan J, Chen A, Rabadan R, Schwartz GK. A Phase I Study of the Combination of Pexidartinib and Sirolimus to Target Tumor-Associated Macrophages in Unresectable Sarcoma and Malignant Peripheral Nerve Sheath Tumors. Clin Cancer Res. 2021 Oct 15;27(20):5519-5527. doi: 10.1158/1078-0432.CCR-21-1779. Epub 2021 Jul 28. PMID 34321280
- See also: Herbert Irving Comprehensive Cancer Center — http://www.hiccc.columbia.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1, Phase 1: Subjects with unresectable or metastatic sarcoma will take orally 800 mg pexidartinib in combination with 2 mg sirolimus daily (Dose Level 2).
- Cohort 2, Phase 1: Subjects with unresectable or metastatic sarcoma will take orally 1000 mg pexidartinib in combination with 2 mg sirolimus daily (Dose Level 3).
- Cohort 3, Phase 1: Subjects with unresectable or metastatic sarcoma will take orally 1000 mg pexidartinib in combination with 4 mg sirolimus daily (Dose Level 4).
- Cohort 4, Phase 1: Subjects with unresectable or metastatic sarcoma will take orally 1000 mg pexidartinib in combination with 6 mg sirolimus daily (Dose Level 5).
- Phase 2 Cohort: Subjects with unresectable or metastatic Malignant Peripheral Nerve Sheath Tumors (MPNSTs) will take the recommended Phase 2 dose (RP2D): 1000 mg pexidartinib and 2 mg sirolimus daily.
Period: Dose Level 1 (S: 2mg, P: 600mg)
Arm/Group | Cohort 1, Phase 1 | Cohort 2, Phase 1 | Cohort 3, Phase 1 | Cohort 4, Phase 1 | Phase 2 Cohort
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2 (S: 2mg, P:800mg)
Arm/Group | Cohort 1, Phase 1 | Cohort 2, Phase 1 | Cohort 3, Phase 1 | Cohort 4, Phase 1 | Phase 2 Cohort
Started | 2 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Level 3 (S: 2mg, P: 1000mg)
Arm/Group | Cohort 1, Phase 1 | Cohort 2, Phase 1 | Cohort 3, Phase 1 | Cohort 4, Phase 1 | Phase 2 Cohort
Started | 0 | 12 | 0 | 0 | 0
Completed | 0 | 9 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 0
Period: Dose Level 4 (S: 4mg, P: 1000mg)
Arm/Group | Cohort 1, Phase 1 | Cohort 2, Phase 1 | Cohort 3, Phase 1 | Cohort 4, Phase 1 | Phase 2 Cohort
Started | 0 | 0 | 9 | 0 | 0
Completed | 0 | 0 | 6 | 0 | 0
Not Completed | 0 | 0 | 3 | 0 | 0
Period: Dose Level 5 (S: 6mg, P: 1000mg)
Arm/Group | Cohort 1, Phase 1 | Cohort 2, Phase 1 | Cohort 3, Phase 1 | Cohort 4, Phase 1 | Phase 2 Cohort
Started | 0 | 0 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: RP2D (S: 2mg, P: 1000mg)
Arm/Group | Cohort 1, Phase 1 | Cohort 2, Phase 1 | Cohort 3, Phase 1 | Cohort 4, Phase 1 | Phase 2 Cohort
Started | 0 | 0 | 0 | 0 | 14
Completed | 0 | 0 | 0 | 0 | 14
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1, Phase 1 | Cohort 2, Phase 1 | Cohort 3, Phase 1 | Cohort 4, Phase 1 | Phase 2 Cohort | Total
Number analyzed (Participants) | 2 | 12 | 9 | 1 | 14 | 38
Age, Continuous [Median (Full Range); unit: years] | 52.5 [52 to 53] | 47.0 [22 to 70] | 60 [21 to 72] | 44 [44 to 44] | 36.5 [19 to 72] | 49.4 [19 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 2 | 1 | 4 | 16
  Male | 1 | 4 | 7 | 0 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 1 | 2 | 6
  Not Hispanic or Latino | 1 | 10 | 9 | 0 | 12 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 1 | 0 | 1 | 5
  White | 1 | 6 | 7 | 0 | 12 | 26
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 0 | 1 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 12 | 9 | 1 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) - Phase 1
Description: The highest dose of a drug or treatment that does not cause unacceptable side effects, which will be used in Phase 2.
Time Frame: Up to 3 years
Measure: Number; unit: mg
Groups:
- Phase 1: Subjects with unresectable or metastatic sarcoma will take orally PLX3397 (600 - 1000mg) in combination with Sirolimus (2-6mg) daily during Phase 1 of the study.
Arm/Group | Phase 1
Number analyzed (Participants) | 24
mg
  Pexidartinib | 1000
  Sirolimus | 2

2. Primary Outcome: Progression Free Survival (PFS) Rate - Phase 2
Description: The time from the start of treatment until disease progression or death from any cause, calculated in weeks.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- Phase 2: Subjects with unresectable or metastatic Malignant Peripheral Nerve Sheath Tumors (MPNSTs) will take the recommended Phase 2 dose (RP2D): 1000 mg pexidartinib and 2 mg sirolimus daily.
Arm/Group | Phase 2
Number analyzed (Participants) | 14
weeks | 6 [6 to 19.1]

3. Secondary Outcome: Overall Survival Rate
Description: The time from the start of treatment until death, estimated using the Kaplan Meier method.
Time Frame: Up to 3 years
Population: Only assessed for Phase 2
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2
Number analyzed (Participants) | 14
weeks | 17.9 [13.7 to NA] — insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Up to 4 years
Groups:
- Cohort 1, Phase 1: Subjects with unresectable or metastatic sarcoma will take orally 800 mg pexidartinib in combination with 2 mg sirolimus daily.
- Cohort 2, Phase 1: Subjects with unresectable or metastatic sarcoma will take orally 1000 mg pexidartinib in combination with 2 mg sirolimus daily.
- Cohort 3, Phase 1: Subjects with unresectable or metastatic sarcoma will take orally 1000 mg pexidartinib in combination with 4 mg sirolimus daily.
- Cohort 4, Phase 1: Subjects with unresectable or metastatic sarcoma will take orally 1000 mg pexidartinib in combination with 6 mg sirolimus daily.
- Phase 2 Cohort: Subjects with unresectable or metastatic Malignant Peripheral Nerve Sheath Tumors (MPNSTs) will take pexidartinib and sirolimus at the recommended Phase 2 dose (RP2D): 1000 mg pexidartinib in combination with 2 mg sirolimus daily.
Arm/Group | Cohort 1, Phase 1 | Cohort 2, Phase 1 | Cohort 3, Phase 1 | Cohort 4, Phase 1 | Phase 2 Cohort
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/12 | 1/9 | 0/1 | 1/14
Serious Adverse Events (participants affected / at risk) | 1/2 | 6/12 | 7/9 | 0/1 | 5/14
Other Adverse Events (participants affected / at risk) | 2/2 | 12/12 | 9/9 | 1/1 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Phase 1 (N=2) | Cohort 2, Phase 1 (N=12) | Cohort 3, Phase 1 (N=9) | Cohort 4, Phase 1 (N=1) | Phase 2 Cohort (N=14)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | NA | 0
Social circumstances (Social circumstances) | 0 | 1 | 0 | NA | 0
Sepsis (Immune system disorders) | 0 | 1 | 0 | NA | 0
Pain (General disorders) | 0 | 1 | 1 | NA | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | NA | 0
Dehydration (General disorders) | 0 | 1 | 0 | NA | 0
Vomiting (General disorders) | 0 | 1 | 1 | NA | 0
Nervous system disorders (Nervous system disorders) | 0 | 1 | 0 | NA | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 1
Hyperkalemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | NA | 0
Administration site condition (General disorders) | 0 | 0 | 1 | NA | 0
Nausea (General disorders) | 0 | 0 | 1 | NA | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | NA | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | NA | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | NA | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 0 | 1 | NA | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | NA | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | NA | 1
Syncope (General disorders) | 0 | 0 | 0 | NA | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1, Phase 1 (N=2) | Cohort 2, Phase 1 (N=12) | Cohort 3, Phase 1 (N=9) | Cohort 4, Phase 1 (N=1) | Phase 2 Cohort (N=14)
Alanine aminotransferase increased (Hepatobiliary disorders) | 2 | 3 | 2 | 1 | 3
Alkaline phosphatase increased (Hepatobiliary disorders) | 2 | 4 | 4 | 1 | 3
Allergic rhinitis (General disorders) | 0 | 0 | 1 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 10 | 5 | 1 | 3
Anorexia (General disorders) | 0 | 5 | 6 | 1 | 6
Anxiety (General disorders) | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (General disorders) | 2 | 9 | 5 | 1 | 3
Bloating (General disorders) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0
Blurred vision (General disorders) | 0 | 0 | 1 | 1 | 0
Bruising (General disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 2 | 0 | 0
Confusion (General disorders) | 0 | 1 | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 4 | 4 | 0 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 0 | 2
Creatinine increased (General disorders) | 2 | 4 | 4 | 0 | 0
Dehydration (General disorders) | 0 | 1 | 1 | 0 | 0
Depression (General disorders) | 0 | 0 | 1 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 4 | 4 | 0 | 6
Dry mouth (General disorders) | 0 | 0 | 2 | 0 | 0
Dysgeusia (General disorders) | 0 | 4 | 3 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4 | 1 | 2
Edema (General disorders) | 0 | 1 | 3 | 0 | 2
Epistaxis (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 7 | 7 | 1 | 6
Fever (General disorders) | 0 | 2 | 3 | 0 | 2
Hallucinations (General disorders) | 0 | 1 | 0 | 0 | 0
Headache (General disorders) | 1 | 0 | 1 | 1 | 0
Hematoma (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 2 | 0 | 2
Hypercalcemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0
Hyperglycemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Hyperkalemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1
Hypernatremia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Hypertension (General disorders) | 1 | 3 | 1 | 1 | 1
Hyperuricemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0
Hypoalbuminemia (Blood and lymphatic system disorders) | 0 | 3 | 4 | 0 | 0
Hypocalcemia (Blood and lymphatic system disorders) | 0 | 4 | 5 | 1 | 0
Hypoglycemia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 0
Hypokalemia (Blood and lymphatic system disorders) | 0 | 4 | 4 | 0 | 3
Hyponatremia (Blood and lymphatic system disorders) | 0 | 4 | 3 | 0 | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0
Hypoxia (General disorders) | 0 | 0 | 1 | 0 | 0
INR increased (Blood and lymphatic system disorders) | 0 | 4 | 3 | 1 | 0
Insomnia (General disorders) | 0 | 1 | 0 | 1 | 2
Laryngeal hemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Lip infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 | 5 | 5 | 1 | 2
Mucositis oral (General disorders) | 0 | 2 | 1 | 0 | 0
Nasal congestion (General disorders) | 1 | 0 | 0 | 0 | 0
Nausea (General disorders) | 0 | 6 | 6 | 1 | 4
Nervous system disorders (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Immune system disorders) | 0 | 4 | 1 | 1 | 6
Oral dysesthesia (General disorders) | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 2 | 7 | 3 | 1 | 12
Paresthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 0 | 2 | 4 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 3 | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 5 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (General disorders) | 0 | 1 | 2 | 0 | 0
Weight loss (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 0
White blood cell decreased (Blood and lymphatic system disorders) | 0 | 5 | 3 | 0 | 4

LIMITATIONS AND CAVEATS:
In the present study, the combination of pexidartinib and sirolimus failed to meet the primary endpoint in a study that was stopped due to poor enrollment due to COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT02584647/Prot_SAP_000.pdf